CLINICAL TRIAL: NCT07334301
Title: A Multi-Arm, Multi-Stage Platform Trial For Relapsed Neuroblastoma
Brief Title: A Multi-Arm, Platform Trial For Relapsed Neuroblastoma
Acronym: BEACON2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_22-136
Record Dates: First submitted 2025-09-12; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Neuroblastoma
Keywords: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Bevacizumab; dinutuximab; Irinotecan; Pharmaceutical Preparations; Topotecan; Temozolomide

STUDY DESIGN:
Intervention Model Description: Multi Arm Multi Stage (MAMS) design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: dinutuximab, irinotecan and temozolomide (dbIT) (Active Comparator)
  Interventions: Drug: Dinutuximab beta; Drug: Irinotecan (drug); Drug: Topotecan; Drug: Temozolomide (TMZ)
- Arm B: bevacizumab, irinotecan and temozolomide (BIT) (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Irinotecan (drug); Drug: Topotecan; Drug: Temozolomide (TMZ)
- Arm C: dinutuximab, bevacizumab, irinotecan and temozolomide (dbBIT) (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Dinutuximab beta; Drug: Irinotecan (drug); Drug: Topotecan; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab
  Arms: Arm B: bevacizumab, irinotecan and temozolomide (BIT); Arm C: dinutuximab, bevacizumab, irinotecan and temozolomide (dbBIT)
Drug: Dinutuximab beta — Dinutuximab beta
  Arms: Arm A: dinutuximab, irinotecan and temozolomide (dbIT); Arm C: dinutuximab, bevacizumab, irinotecan and temozolomide (dbBIT)
Drug: Irinotecan (drug) — Irinotecan
Drug: Topotecan — Topotecan
Drug: Temozolomide (TMZ) — Temozolomide capsule
Drug: Temozolomide (TMZ) — Temozolomide liquid suspension

SUMMARY:
Neuroblastoma is one of the most common solid childhood tumours, and a major cause of cancer-related death in children. More than 1200 children/young adults a year are diagnosed in USA and Europe. Around 600 of these cases are considered high-risk, which means the cancer is more difficult to treat successfully. Despite improvements in survival over recent decades, a significant proportion of patients with high-risk neuroblastoma have disease that does not respond to standard treatments (refractory neuroblastoma) or comes back after completion of standard frontline treatment (relapsed neuroblastoma). Therefore, there is a need to develop new treatment strategies and test new drugs to improve outcomes for children with neuroblastoma.

Aims Of The BEACON2 Trial

* To improve survival for patients with relapsed neuroblastoma by developing new treatment combinations
* To evaluate new treatment combinations in relapsed neuroblastoma, within a phase I/II trial that can impact clinical practice, while also allowing dose confirmation for new promising combinations
* To evaluate the safety, activity, efficacy and impact on quality of life of these new treatment combinations in relapsed neuroblastoma patients
* To improve our understanding of relapsed neuroblastoma biology and advance the development of targeted therapies using biomarkers, by conducting a comprehensive biomarker sample collection.

Trial Design BEACON2 is a randomised phase I/phase II, open label, international trial. The trial will have two tiers: Tier 1 will be the main randomisation for two treatment arms initially. Participants will be randomised at trial entry to receive one of the available regimens, treatment A or treatment B. Tier 2 will include smaller dose expansion/confirmation cohorts for more novel experimental treatment combinations (Arm C and future arms), with the potential for them to be moved to Tier 1.

Current Tier 1 (Randomisation Tier) Treatment Arms in the BEACON2 Trial:

Arm A: dbIT Treatment with dinutuximab beta, irinotecan, and temozolomide, 3 weekly x12 cycles Arm B: BIT Treatment with bevacizumab, irinotecan, and temozolomide, 3 weekly x12 cycles

Current Tier 2 (Registration Only Tier) Treatment Arms in the BEACON2 Trial:

Arm C: dbBIT Treatment with dinutuximab beta, bevacizumab, irinotecan, and temozolomide, 3 weekly x12 cycles

Patient Population and Sample Size Patients aged ≥1 years of age with relapsed neuroblastoma. For each arm in Tier 1, up to 75 patients will be recruited to complete phase 2 investigations. For each arm in Tier 2, 10 patients will be recruited to complete phase I investigations. Approximately 160 participants are initially planned, 75 in each arm of Tier 1 and 10 participants for one dose-confirmation cohort in Tier 2.

The study is expected to recruit patients for 3 years, and then finish patient follow-up after an additional 5 years.

Translational Sub-study / Biological Studies

It is standard of care for patients diagnosed with relapsed neuroblastoma to:

* Have had a tumour sample collected at point of initial diagnosis (either during biopsy or surgery)
* Have bloods collected before they start and during treatment for their relapsed neuroblastoma
* Have a bone aspirate/trephine procedure in order to help confirm relapse. These samples provide very important opportunities for further research, and the study investigators would like to make full use of these opportunities by collecting the analysis already performed on these samples and collect some additional samples (at the same time as the standard ones) to learn and understand more about neuroblastoma and its treatment. Samples will undergo research analysis at the national SIOPEN reference laboratories.

ELIGIBILITY:
Inclusion Criteria:

* Disease specific

  * Histologically proven neuroblastoma as per International Neuroblastoma Staging System (INSS)[1] definition
  * High risk relapsed neuroblastoma (relapsed or progressed after being defined as High Risk at any time following diagnosis or progressed/relapsed as high-risk neuroblastoma)
  * Measurable disease by cross sectional imaging or evaluable disease (uptake on MIBG scan with or without bone marrow histology), as per INRC [2, 3]. Participants with only bone marrow detectable disease (bone marrow aspirate or trephine) are NOT eligible for the study General
  * Age ≥1 year
  * Signed informed consent from participant, parent or guardian Performance and organ function
  * Performance Status

    o Lansky (for patients ≤12 years of age) or Karnofsky (for those >12) ≥ 50%, (Participants who are unable to walk because of paralysis, but who are able to sit upright unassisted in a wheelchair, will be considered ambulatory for the purpose of assessing performance score)
  * Life expectancy of ≥12 weeks
  * Bone marrow function (within 72 hours prior to randomisation):

    * Platelets ≥ 50 x 109/L (unsupported for 72 hours)
    * ANC ≥ 0.50 x 109/L (no G-CSF support for 72 hours)
    * Haemoglobin > 8 g/dL (transfusions allowed)
  * Renal function (within 72 hours prior to randomisation):

    * Absence of clinically significant proteinuria (either early morning urine dipstick ≤ 2+) or if dipstick urinalysis shows > 2+ proteinuria, protein: creatinine (Pr/Cr) ratio must be < 0.5 or a 24 hour protein excretion must be < 0.5g
    * Serum creatinine ≤ 1.5 ULN for age, if higher, a measured GFR (radioisotope or 24 hour urine calculated creatinine clearance) must be ≥ 60 ml/min/1.73 m2
  * Liver function (within 72 hours prior to randomisation):

    o Absence of clinically significant signs of liver dysfunction. AST or ALT ≤ 3.0 ULN and total bilirubin ≤ 1.5 ULN. In patients with liver metastases, AST or ALT ≤ 5 ULN and total bilirubin ≤ 2.5 ULN is allowed.
  * Coagulation:

    * Participants must not have an active uncontrolled coagulopathy.
    * Anticoagulation is permitted as long as the INR or APTT is within therapeutic limits (according to the medical standard of the institution) and the participant has been on a stable dose of anticoagulants for at least two weeks at the time of study enrolment.
  * Blood pressure below 95th centile for age and sex. Participants ≥18 years of age should have a blood pressure ≤150/90 mmHg (within 72 hours prior to randomisation). Use of antihypertensive medication is permitted.

Tier 2 Specific Inclusion Criteria

• More than one relapse event or ineligible for Tier 1.

NB- The following previous treatments are allowed provided that the principal investigator expects a favourable benefit/risk assessment (e.g. patients could derive potential benefit from the Tier 2 combination):

* bevacizumab,
* any anti-GD2 antibody given with chemotherapy ('chemo-immunotherapy')
* previous treatment with temozolomide with irinotecan

Exclusion Criteria:

* • Known contraindication or hypersensitivity to:

  * Any study drug or component of the formulation
  * Chinese hamster ovary products or other recombinant human or humanised antibodies.
  * Participants with mild previous hypersensitivity reactions to anti-GD2 antibodies may be included, but those with severe (or G4) hypersensitivity reactions to anti-GD2 antibodies will be excluded.

    * Clinically significant neurological toxicity, uncontrolled seizures or objective peripheral neuropathy (> grade 2). (Unresolved neurological deficits from previous spinal cord compression or surgeries are acceptable). Participants with previous ≥ Grade 3 motor neurotoxicity secondary to anti-GD2 are excluded, even if recovered
    * Prior severe arterial thrombo-embolic events (e.g. cardiac ischemia, cerebral vascular accident, peripheral arterial thrombosis) or any ongoing arterial thrombo-embolic events
    * A history of (noninfectious) pneumonitis requiring steroids, or current pneumonitis.
    * Patients that are allergic to all therapies for Pnemocystis jirovecii pneumonia and can thus not receive prophylaxis for PJP
    * Uncontrolled infection
    * Inadequate recovery from prior surgery with ongoing ≥ Grade 3 surgical complications. Grade ≥ 2 wound dehiscence.
    * Recent surgical procedures (at start of trial treatment). Patient can be randomised up to 48hr prior to these periods being completed provided that trial treatment only starts after complying with all of them:
  * Core biopsies within previous 24hr
  * Open excisional biopsies within previous 48hr
  * Major surgery within previous 2 weeks
  * Bone marrow aspirates/trephines, within previous 48hr
  * Tunnelled central line insertion within previous 48hr

    • Washout from prior treatments (at start of trial treatment):
  * Chemotherapy within previous 2 weeks (1 week for oral metronomic chemotherapy regimens)
  * Any anti-GD2 therapy within previous 2 weeks
  * Craniospinal radiotherapy or MIBG therapy within previous 6 weeks
  * Radiotherapy to the tumour bed within previous 2 weeks (no washout for palliative radiotherapy)
  * Myeloablative therapy with haematopoietic stem cell rescue (autologous stem cell transplant) within previous 8 weeks
  * Allogeneic stem cell transplant within previous 12 weeks (with absence of active ≥ G2 acute GVHD)
  * 14 days or 5 half-lives (whichever occurs later) from last administration of an IMP in an IMP-trial

    * Bleeding metastases (participants with CNS metastases can be enrolled as long as the metastases are not bleeding). At least 6 months from any ≥ G3 haemoptysis or pulmonary haemorrhage
    * Use of enzyme inducing anticonvulsants within 72hr of start of trial treatment
    * Conditions that increase the risk of bevacizumab-related toxicities:
  * History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e. in the absence of therapeutic anticoagulation)
  * History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or active gastrointestinal bleeding within 6 months prior to study enrolment
  * Current chronic intestinal inflammatory disease/bowel obstruction

    * Intolerance to galactose and fructose, lactase deficiency, and/or defect of absorption of galactose and fructose
    * Males or females of reproductive potential may not participate unless they agree to use a highly effective method of birth control, i.e. with a failure rate of less than 1% per year, (e.g. implants, injectables, combined oral contraceptives, IUDs, sexual abstinence or vasectomised partner), for the duration of study therapy and for up to 6 months after the last dose of trial drugs. A negative urine or serum pregnancy test must be obtained within 72 hours prior to dosing in females who are post-menarche.
    * Pregnant or lactating participant
    * Live or live-attenuated vaccines given within previous 28 days prior to study enrolment
    * Any uncontrolled medical condition that poses an additional risk to the participant

Tier 1 Specific Exclusion Criteria

* More than one relapse/progression event after the start of high risk neuroblastoma therapy
* Previous treatments that are not allowed

  * Bevacizumab for relapsed neuroblastoma. Patients who have received BIT for refractory disease are not excluded, providing no progression of disease during this treatment occurred
  * Treatment with any anti-GD2 antibody given with chemotherapy ('chemo-immunotherapy') for treatment of relapsed neuroblastoma. Prior treatment with chemo-immunotherapy for refractory disease is allowed, provided no disease progression during this therapy.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival time | From date of randomization until the date of first documented failure event (progression or death), assessed up to 60 months.
  • Progression-Free Survival time (as per International Neuroblastoma Response Criteria (PD Progressive disease, SD Stable disease, MR Minor response, PR Partial response, CR Complete response) INRC 2017) - for Tier 1 (randomised comparison)
Occurrence of dose-limiting toxicities to definition of a safe and tolerable combination regimen | From date of randomization until the date of first documented failure event (progression or death), assessed up to 60 months.
  Tier 2 (dose expansion-confirmation cohorts): Definition of a safe and tolerable (i.e. </= 3 dose-limiting toxicities) combination regimen

SECONDARY OUTCOMES:
Best objective response | At the end of the last treatment cycle, up to 12 cycles (each cycle is 21 days)
  Best objective response (complete and partial response) per the INRC 2017 during trial treatment (12 cycles)
Clinical benefit | At the end of the last treatment cycle, up to 12 cycles (each cycle is 21 days)
  Clinical benefit (complete, partial and minor response and stable disease) per the INRC 2017 (International Neuroblastoma Response Criteria (PD Progressive disease, SD Stable disease, MR Minor response, PR Partial response, CR Complete response))
Time response to progression | From date of response (Complete Response, Partial Response or Minor Response as per INRC) until the date of first documented failure event (progression or death), assessed up to 60 months.
  Time between Response to Progression (i.e. Duration of Response) for patients who respond
Overall Survival time | From date of trial entry until the date of first documented failure event (progression or death), assessed up to 60 months.
  Overall Survival time
Quality of life of patients measured by Peds-QL questionnaires | At the end of the last treatment cycle, up to 12 cycles (each cycle is 21 days)
  Quality of life of patients measured by Pediatric Quality of Life Inventory (Peds-QL) questionnaires. 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher PedsQL 3.0 scores indicate better Health Related Quality of Life (HRQOL).
Incidence and Severity of AEs | From date of trial entry until the date of last follow up, assessed up to 60 months.
  Incidence and Severity of AEs

OTHER OUTCOMES:
Quality of life of caregivers measured by Peds-QL questionnaires | At the end of the last treatment cycle, up to 12 cycles (each cycle is 21 days)
  Quality of life of caregivers measured by Pediatric Quality of Life Inventory (Peds-QL) questionnaires. 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher PedsQL 3.0 scores indicate better Health Related Quality of Life (HRQOL)
Correlation between objective response using INRC 2017 and PFS/OS | At the end of the last treatment cycle, up to 12 cycles (each cycle is 21 days)
  Correlation between objective response using INRC 2017 and PFS/OS
Changes in circulating biomarkers and tumour molecular profiles in tumour and blood | At the end of the last treatment cycle, up to 12 cycles (each cycle is 21 days)
  Changes molecular and genetic profile of tumour and blood as measured by genetic analysis at baseline and throughout the study.

CONTACTS AND LOCATIONS:
Locations (23):
- Sydney Children's Hospital (SCH), Sydney, Australia
- St. Anna Children´s Hospital, Vienna, Austria
- Cliniques Universitaires Saint-Luc (CUSL), Brussels, Belgium
- Starship Children's Hospital (SSH), Auckland, New Zealand
- United Kingdom (19):
  - Royal Aberdeen Children's Hospital, Aberdeen
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrookes Hospital, Cambridge
  - Children's Hospital for Wales, Cardiff
  - Royal Hospital for Sick Children, Edinburgh
  - Royal Hospital for Children, Glasgow
  - Leeds General Infirmary, Leeds
  - Alder Hey Hospital, Liverpool
  - Great Ormond Street Hospital, London
  - University College London Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham Children's Hospital, Nottingham
  - John Radcliffe Hospital, Oxford
  - Sheffield Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brodeur GM, Pritchard J, Berthold F, Carlsen NL, Castel V, Castelberry RP, De Bernardi B, Evans AE, Favrot M, Hedborg F, et al. Revisions of the international criteria for neuroblastoma diagnosis, staging, and response to treatment. J Clin Oncol. 1993 Aug;11(8):1466-77. doi: 10.1200/JCO.1993.11.8.1466. PMID 8336186

DOCUMENTS (1):
  • Study Protocol (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT07334301/Prot_000.pdf